CLINICAL TRIAL: NCT04868422
Title: Wireless Telemonitoring of Nasal CPAP Therapy in Sleep Apnea Patients
Brief Title: Telemonitoring of CPAP Therapy in Sleep Apnea Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Tarja Saaresranta, Investigator, University of Turku
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T83/2012; K53 (Other: Turku University Hospital)
Record Dates: First submitted 2021-04-26; First posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: sleep apnea; CPAP treatment; telemedicine; nursing time; patient satisfaction
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: The Ethics Committee approval was not required, since this study was part of our quality assurance procedure to revise the treatment protocol.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemonitoring (Experimental): After CPAP titration, patients will be followed with telemonitoring device attached to the fixed pressure CPAP device
  Interventions: Device: Telemonitoring via wireless internet-based system
- Usual care (No Intervention): Patients with fixed pressure CPAP will be followed according to routine protocol without telemonitoring

INTERVENTIONS:
Device: Telemonitoring via wireless internet-based system
  Arms: Telemonitoring

SUMMARY:
Wireless telemonitoring is compared with regular nursing procedure in terms of patient satisfaction, adherence to continuous positive pressure (CPAP) treatment and nursing time during the habituation phase of the CPAP therapy in obstructive sleep apnea syndrome (OSAS).

DETAILED DESCRIPTION:
Both patients and study nurses were unblinded for the wireless telemonitoring system (ResTraxx™Online, ResMed, Sydney, Australia). The module was attached to the S9 Elite™ (ResMed, Sydney, Australia) CPAP device, which transmitted compliance data every day automatically to the ResTraxx™ Online (ResMed, Sydney, Australia) data base. The treatment was considered successful when CPAP use was >4 h/day, mask leak <0.4 L/s, and AHI <5/h during the last 6 days. Study nurses made the data check-ups daily during weekdays and if the criteria for successful CPAP therapy was not achieved during two consecutive nights the nurses adjusted the CPAP pressure remotely and called the patient to give further advice. Patients had also a control viist aftr one year.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with diagnosed obstructive sleep apnea

Exclusion Criteria:

* Not able to understand Finnish language
* Unable to co-operate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2012-08-14 (Actual); Primary Completion 2014-08-12 (Actual); Study Completion 2015-03-12 (Actual)

PRIMARY OUTCOMES:
Nursing time | One year after the baseline
  Nursing time of the TM group was estimated as follows: patient education regarding ResTraxx™ Online system (2 min), online data check-ups (0.5 min), remote changes for pressure settings (1 min), telephone guidance (5 min for the end of monitoring, 10 min for each extra call), visit at the study nurse (30- 60 min depending on type of visit), updating the patient records (2 min), and no show visits, which led to organizing a new appointment (20min). The time estimations are based on the measurements of the first 20 telemonitored patients. Nursing time in the UC Group was estimated with the same time calculations as in the TM group presented above with the exception of ttelemonitoring time which was not applicable in the UC group.

SECONDARY OUTCOMES:
Hours of CPAP use | One year after baseline
  Hours of CPAP use measured by the inbuilt counter of the CPAP device

OTHER OUTCOMES:
Residual apnea-hypopnea index (AHI) | One year after baseline
  Maan AHI over 12 months according the CPAP-device

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital, Turku, Finland